CLINICAL TRIAL: NCT02677233
Title: Association Between Vitamin D Deficiency and Preeclampsia: A Case Control Study
Status: Completed | Type: Observational
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Salah sayed, mohamed salah, Ain Shams Maternity Hospital
Other Study IDs: vid-20
Record Dates: First submitted 2016-02-05; First posted 2016-02-09 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- preeclamptic group: 1. Blood pressure: greater than or equal to 140 mmHg systolic or greater than or equal to 90 mmHg diastolic on two occasions at least 4 hours apart after 20 weeks of gestation (Roberts et al., 2013).
  2. Proteinuria: protein/creatinine ratio greater than or equal to 0.3
  3. In the absence of proteinuria, a new-onset hypertension with new onset of the following:
     * thrombocytopenia: platelet count less than 100.000/microliter
     * renal insufficiency: serum creatinine greater than 1.1 mg/dl
     * impaired liver function: elevated concentration of liver transaminases
     * pulmonary edema
     * cerebral or visual symptoms
     * Severe right upper quadrant or epigastric pain unresponsive to medication.
- non preeclamptic group: All are normotensive with blood pressure <140/90 with no proteinuria.

SUMMARY:
To find out if lower levels of vitamin D is more prevalent in preeclamptic women

ELIGIBILITY:
Inclusion Criteria:

* Parity: primigravida.
* Age: 18 - 35 years.
* Singleton pregnancy.
* Gestational age: 36-40 weeks.
* No past history of any medical disorder and with no other medical complications during pregnancy

Exclusion Criteria:

* Women with preexisting medical conditions like rheumatoid arthritis, thyroid, hepatic or renal failure, metabolic bone disease, diabetes mellitus, malabsorption and lupus.
* History of intake of medications influencing bone, vitamin D or calcium metabolism e.g. antiepileptic, theophylline, antitubercular drugs in the last 6 months.
* Women with multiple pregnancy.
* Women with congenital fetal malformation.
* Women with known thrombophilia

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study will be carried out on 90 pregnant women recruited at pre labour room at Ain Shams University Maternity Hospital. They will be divided into preeclamptic group and non preeclamptic group, 45 cases in each one
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
vitamin D level in preeclamptic and non preeclamptic women | six months

IPD SHARING:
Plan to Share IPD: No